CLINICAL TRIAL: NCT03601676
Title: Increasing Safe Outpatient Care for Emergency Department Patients With Acute Pulmonary Embolism: a Pragmatic Trial
Brief Title: Electronic Support for Pulmonary Embolism Emergency Disposition
Acronym: eSPEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CN-13-1738-H
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Pragmatic clinical trial of a multidimensional technology and educational intervention undertaken over 16 months with an 8-month pre-intervention and an 8-month post-intervention period, conducted across 21 emergency departments with 10 serving as intervention and 11 as control sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Other: Integration of electronic clinical decision support
- Control (No Intervention)

INTERVENTIONS:
Other: Integration of electronic clinical decision support — Integration of an electronic clinical decision support system into the emergency department patient care workflow to assist with site-of-care decision-making for emergency department patients with acute pulmonary embolism.
  Arms: Intervention

SUMMARY:
To evaluate the impact of an integrated electronic clinical decision support system to facilitate risk stratification and site-of-care decision-making for patients with acute pulmonary embolism.

DETAILED DESCRIPTION:
Many low-risk emergency department patients with acute pulmonary embolism are routinely hospitalized despite being eligible for outpatient care. One impediment to home discharge is the difficulty of identifying which patients can safely forego hospitalization. This pragmatic clinical trial intends to evaluate the effect on emergency department disposition of a multicomponent intervention, including electronic clinical decision support system access, physician education, and physician-specific audit and feedback. The hypothesis for this study is that intervention sites, when compared with concurrent control sites, will see an increase in home discharges without an increase in 5-day pulmonary embolism-related return visits or 30-day all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Acute objectively-confirmed pulmonary embolism, diagnosed in the emergency department

Exclusion Criteria:

* Comfort-care only
* Left the ED against medical advice
* Current PE radiologically diagnosed >12 hrs prior to arrival
* Recent DVT or PE diagnosed within 30 days
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1703 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Rate of home discharge from the emergency department following treatment for pulmonary embolism | 8 months post-implementation compared to 8 months pre-implementation

SECONDARY OUTCOMES:
Number of participants with major hemorrhage, recurrent venous thromboembolism, and all-cause mortality | 30 days
Number of participants with return visits for pulmonary embolism-related signs, symptoms, or interventions | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: David R Vinson, MD, Principal Investigator — Kaiser Permanente
Locations (14):
- United States (14):
  - Kaiser Permanente Fremont Emergency Department, Fremont, California
  - Kaiser Permanente Oakland Emergency Department, Oakland, California
  - Kaiser Permanente Redwood City Emergency Department, Redwood City, California
  - Kaiser Permanente Richmond Emergency Department, Richmond, California
  - Kaiser Permanente Roseville Emergency Department, Roseville, California
  - Kaiser Permanente South Sacramento Emergency Department, Sacramento, California
  - Kaiser Permanente Sacramento Emergency Department, Sacramento, California
  - Kaiser Permanente San Francisco Emergency Department, San Francisco, California
  - Kaiser Permanente San Jose Emergency Department, San Jose, California
  - Kaiser Permanente San Leandro Emergency Department, San Leandro, California
  - Kaiser Permanente San Rafael Emergency Department, San Rafael, California
  - Kaiser Permanente Santa Clara Emergency Department, Santa Clara, California
  - Kaiser Permanente Santa Rosa Emergency Department, Santa Rosa, California
  - Kaiser Permanente South San Francisco Emergency Department, South San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vinson DR, Mark DG, Chettipally UK, Huang J, Rauchwerger AS, Reed ME, Lin JS, Kene MV, Wang DH, Sax DR, Pleshakov TS, McLachlan ID, Yamin CK, Elms AR, Iskin HR, Vemula R, Yealy DM, Ballard DW; eSPEED Investigators of the KP CREST Network. Increasing Safe Outpatient Management of Emergency Department Patients With Pulmonary Embolism: A Controlled Pragmatic Trial. Ann Intern Med. 2018 Dec 18;169(12):855-865. doi: 10.7326/M18-1206. Epub 2018 Nov 13. PMID 30422263